CLINICAL TRIAL: NCT04827628
Title: Effect of Oryza Sativa l Extract to Serum Lipopolysaccharide, Tight Junction Protein 1 (ZO-1), and Intestinal Microbiota Expression Among Obese Individual
Brief Title: Effect of Oryza Sativa l Extract to LPS, ZO-1, and Intestinal Microbiota in Obese Individuals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hasanuddin University (Other)
Responsible Party: Principal Investigator, Bumi Herman, Assistant Lecturer, Hasanuddin University
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1803211718
Record Dates: First submitted 2021-03-30; First posted 2021-04-01 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Obesity
Keywords: Lipopolysaccharide; Zonula Occludens 1; Obesity; Oryza sativa; Anthocyanin; Intestinal Microbiota
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: a non-randomized trial is implemented involving three arms consists of an obese group as the intervention and two control groups, people with normal Body Mass Index, and Obese.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: To blind the participant, the mixture is given in the darker bottle, and placebo is given the artificial taste similar to the intervention group. This adjustment also blinds the care provider. The outcome assessor is blinded from the allocation of the group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Obese with Oryza sativa extract (Experimental): The group with a body mass index of more than 25 kg/m2 that receive the Oryza Sativa Extract
  Interventions: Dietary Supplement: Oryza Sativa Extract
- Obese with control (Active Comparator): The group with a body mass index of more than 25 kg/m2 that receive the citric acid and sorbitol mixture
  Interventions: Dietary Supplement: Control
- Normal Body Mass Index (Active Comparator): The group with a body mass index of less than 25 kg/m2 that receive the citric acid and sorbitol mixture
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Oryza Sativa Extract — The product is a suspension of 5.6 gram/100 mL given once daily, contains 71.9%, purple in color, range pH 3-5. Stored in the darker bottle. The frequency of administration is once-daily after the meal.
  Arms: Obese with Oryza sativa extract
Dietary Supplement: Control — citric acid 0.1g/oz and 1% sorbitol mixture, given once daily after meal
  Arms: Normal Body Mass Index; Obese with control

SUMMARY:
Background :

Obesity prevalence rises among adults and leads to morbidity and mortality due to subsequent inflammation pathway activation. This activation is induced by higher lipid consumption which activates the Nuclear factor kappa-light-chain-enhancer of activated B cells (NF-kB) pathway and alters the microbiota profile. The Oryza sativa extract contains anthocyanin which possibly affects the microbiota composition and NF-kb pathway which eventually preserves the protective layer and tight junction of the epithelial cells. Therefore it is important to address the impact of this extract on these parameters.

Objective :

To assess the effect of Oryza sativa extract on microbiota profile (Lactobacillus, Firmicutes, Bacteroides, Bifidobacteria, and Escherichia coli), Lipopolysaccharide/ LPS, and the tight epithelial junction (Zonula Occludens-1) among obese adults.

Method:

A two-arm Quasi-Experimental will be conducted, followed by two repeated measurements, at the baseline and 3 weeks after intervention

Hypothesis:

Oryza sativa extract lowers the LPS level, Firmicutes sp, Bacteroides sp, and increases ZO1 protein, Bifidobacteria, and Lactobacillus sp.

DETAILED DESCRIPTION:
Method:

1. Non Randomized clinical trial with double-blind
2. Participants will be recruited consecutively
3. Matching technique will be applied following several variables adjustment
4. Two-arm of the group participants are the normal group, the obese control group, and the obese intervention group

Sample size calculation:

The difference between two independent means sample size calculation is applied following the elements below:

a. Type 1 error: 10% b. Power: 80% c. Effect Size: 0.9 (based on changes of LPS value) d. Dropout rate: 20% e. Hypothesis: Superiority Trial g. The number of participants per group: 14

Intervention :

1. Extract: Liquid extract of Oryza sativa derived from 10 grams of Oryza sativa fine powder. The powder is mixed with 100 ml ethanol 50% and 0.5 ml of hydrochloric acid (HCl) in 300 C for 2 hours. A supernatant is extracted and evaporated at 35 C and dried and 60 C to remove any dissolving agents. This yields an extract of 624.27 mg.
2. Anthocyanin level is measured using a spectrophotometer where 20 microliters of extract added to 2 mL Potassium Chloride (KCl) (with pH 1.0) and 2 ml Sodium Acetate (NaCH3COO) (pH 4.5). Absorption of 500 nm and 700 nm waves are measured and calculated using the cyanide-3-glucoside calculation where :

anthocyanin level : (absorbance x 449.2 x dilution factor x 1000) / 26.9

Control

a. Active comparator using citric acid and sorbitol mixture

Biological sample:

1. Serum sample preparation :

   Participants should undergo fasting for 12 hours. Blood is drawn from the cubital vein to the plain tube and incubated for 30-45 minutes. Centrifugation of sample is done for 15 minutes with 3000 rotation per minute to yield the serum. The supernatant then extracted and stored at -80 C.
2. Feces primary Polymerase Chain Reaction (PCR) using 100-gram feces. The PCR primer for intestinal microbiota are enlisted below :

   1. Total intestinal microbiota (ACTCCTACGGGAGGCAGCAGT ATTACCGCGGCTGCTGGC),
   2. Firmicutes-Lactobacillus (TACATCCCAACTCCAGAACGAAGCAACAGTACCACGACC)),
   3. Bacteroidetes-Bacteroides fragilis (ATAGCCTTCGAAAGRAAGATCCAGTATCAACTGCAATTTTA),
   4. Actinobacteria-Bifidobacterium (CTCCTGGAAACGGGGTGGGGTGTTCTTCCCGATATCTACA),
   5. Proteobacteria-E.Coli (CATGCCGCGTGTATGAAGAACGGGTAACGTCAATGAGCAAA)

Protection of Human subject according to Helsinki Declaration

1. Participants are allowed to receive the information of research including purpose, possible intervention, and side effects.
2. Possible side effect including :
3. Participants are allowed to withdraw from the study for any reason.

Statistical Analysis Plan

1. Descriptive statistic of the baseline
2. The bivariate analysis between all variables and the outcomes
3. Paired t-test is intended to see the difference between microbiota profile, LPS, and ZO1 within groups
4. The independent-test to measure the difference in microbiota profile, LPS, and ZO1 value between groups
5. Alternative statistical test: Linear mixed model to adjust the fixed and random effects.

ELIGIBILITY:
Inclusion Criteria

1. No consumption of the antioxidant supplement
2. No consumption of prebiotic and probiotic
3. Currently not undergo specific diet

Exclusion Criteria

1. Current smoker
2. Diagnosed with chronic diseases
3. Patients with altered kidney and liver function
4. Unable to participate for any reason

Ages: 18 Years to 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-04-10 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Lipopolysaccharide (LPS) level of Serum | Changes of LPS value from baseline to the last day of intervention (three weeks)
  Measured using Enzyme-Linked Immunosorbent Assay (ELISA)
Microbiota Level in Stool sample | Changes of Microbiota value from baseline to the last day of intervention (three weeks)
  Measured using primary PCR of total microbiota, Firmicutes-Lactobacillus, Bacteroidetes-Bacteroides fragilis, Actinobacteria-Bifidobacterium and Proteobacteria-E.Coli

SECONDARY OUTCOMES:
Zonula Occludens 1 (ZO1) serum level | Changes of ZO1 value from baseline to the last day of intervention (three weeks)
  Measured using Enzyme-Linked Immunosorbent Assay (ELISA)

CONTACTS AND LOCATIONS:
Overall Officials: Agussalim Bukhari, Ph.D, Principal Investigator — Hasanuddin University; Nurpudji Taslim, Prof., Principal Investigator — Hasanuddin University; Aminuddin Aminuddin, Ph.D, Principal Investigator — Hasanuddin University; Armanto Makmun, M.Kes, Principal Investigator — Universitas Muslim Indonesia; Rachmat Syamsu, M.Kes, Principal Investigator — Universitas Muslim Indonesia; Bumi Herman, MD. Ph.D, Principal Investigator — Chulalongkorn University
Locations (1):
- Hasanuddin University Medical Research Center / HUMRC, Makassar, South Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: No
Only protocol could be shared for public

REFERENCES:
- [Background] Aguirre M, Venema K. Does the Gut Microbiota Contribute to Obesity? Going beyond the Gut Feeling. Microorganisms. 2015 Apr 27;3(2):213-35. doi: 10.3390/microorganisms3020213. PMID 27682087
- [Background] Angelakis E, Armougom F, Million M, Raoult D. The relationship between gut microbiota and weight gain in humans. Future Microbiol. 2012 Jan;7(1):91-109. doi: 10.2217/fmb.11.142. PMID 22191449
- [Background] Tehrani AB, Nezami BG, Gewirtz A, Srinivasan S. Obesity and its associated disease: a role for microbiota? Neurogastroenterol Motil. 2012 Apr;24(4):305-11. doi: 10.1111/j.1365-2982.2012.01895.x. Epub 2012 Feb 20. PMID 22339979
- [Background] Tan J, Li Y, Hou DX, Wu S. The Effects and Mechanisms of Cyanidin-3-Glucoside and Its Phenolic Metabolites in Maintaining Intestinal Integrity. Antioxidants (Basel). 2019 Oct 12;8(10):479. doi: 10.3390/antiox8100479. PMID 31614770
- [Background] Morais CA, de Rosso VV, Estadella D, Pisani LP. Anthocyanins as inflammatory modulators and the role of the gut microbiota. J Nutr Biochem. 2016 Jul;33:1-7. doi: 10.1016/j.jnutbio.2015.11.008. Epub 2015 Nov 26. PMID 27260462
- [Background] Min SW, Ryu SN, Kim DH. Anti-inflammatory effects of black rice, cyanidin-3-O-beta-D-glycoside, and its metabolites, cyanidin and protocatechuic acid. Int Immunopharmacol. 2010 Aug;10(8):959-66. doi: 10.1016/j.intimp.2010.05.009. PMID 20669401
- [Background] Lee B, Moon KM, Kim CY. Tight Junction in the Intestinal Epithelium: Its Association with Diseases and Regulation by Phytochemicals. J Immunol Res. 2018 Dec 16;2018:2645465. doi: 10.1155/2018/2645465. eCollection 2018. PMID 30648119
- [Background] Ito VC, Lacerda LG. Black rice (Oryza sativa L.): A review of its historical aspects, chemical composition, nutritional and functional properties, and applications and processing technologies. Food Chem. 2019 Dec 15;301:125304. doi: 10.1016/j.foodchem.2019.125304. Epub 2019 Jul 31. PMID 31394335
- [Background] Igwe EO, Charlton KE, Probst YC, Kent K, Netzel ME. A systematic literature review of the effect of anthocyanins on gut microbiota populations. J Hum Nutr Diet. 2019 Feb;32(1):53-62. doi: 10.1111/jhn.12582. Epub 2018 Jul 8. PMID 29984532
- [Background] Hersoug LG, Moller P, Loft S. Gut microbiota-derived lipopolysaccharide uptake and trafficking to adipose tissue: implications for inflammation and obesity. Obes Rev. 2016 Apr;17(4):297-312. doi: 10.1111/obr.12370. Epub 2015 Dec 29. PMID 26712364
- [Background] Bae IY, An JS, Oh IK, Lee HG. Optimized preparation of anthocyanin-rich extract from black rice and its effects on in vitro digestibility. Food Sci Biotechnol. 2017 Aug 28;26(5):1415-1422. doi: 10.1007/s10068-017-0188-x. eCollection 2017. PMID 30263677